CLINICAL TRIAL: NCT03963791
Title: Remineralization Effect of Eggshell Powder on Post-orthodontic White Spot Lesions Compared to CPP-ACP: A Randomized Controlled Clinical Trial.
Brief Title: Remineralization Effect of Eggshell Powder on Post-orthodontic White Spot Lesions Compared to CPP-ACP
Acronym: REEPP-WSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammad A Sarhan, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oper_607
Record Dates: First submitted 2019-05-15; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Biological Products

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eggshell powder gel (Experimental): prepared from eggshell powder. applied on the tooth surfaces twice daily (after breakfast and before bedtime) after brushing the teeth.
  Interventions: Other: Eggshell powder gel; Other: CPP-ACP crème
- CPP-ACP crème (Active Comparator): CPP-ACP crème (GC Tooth Mousse). applied on the tooth surfaces twice daily (after breakfast and before bedtime) after brushing the teeth.
  Interventions: Other: Eggshell powder gel; Other: CPP-ACP crème

INTERVENTIONS:
Other: Eggshell powder gel — Eggshell powder gel produced from chicken eggs.
  Other Names: Natural product
Other: CPP-ACP crème — A water-based, sugar-free topical cream containing Recaladent (CCP-ACP) which is derived from the milk protein.
  Other Names: MI Paste

SUMMARY:
This research is conducted to compare the remineralization efficacy of eggshell powder gel and CPP-ACP (MI paste) on post-orthodontic white spot lesions.

ELIGIBILITY:
Inclusion Criteria:

* A patient who has just completed a comprehensive orthodontic treatment.
* Presence of at least one WSL, DIAGNOdent score (0-20).
* Age range between 13 and 35years.

Exclusion Criteria:

* Patients are unable to return for recall appointments.
* High caries risk.
* Have plaque accumulation and a periodontal problem
* In progress treatment of chronic disease.
* Presence of abnormal oral, medical, or mental condition (including any milk-related allergies or any medical condition involving kidneys or salivary glands).
* Presence of dentin caries, enamel hypoplasia or restorations on maxillary anterior teeth.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-05 (Estimated); Primary Completion 2020-04-05 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
white spot lesion progression. | 6 months.
  The change in the lesion fluorescence will be evaluated using diode laser fluorescence device (Diagnodent).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo univercity, Cairo, Egypt